CLINICAL TRIAL: NCT03121248
Title: A Partially Randomized Patient Preference Trial, Comparing Adjuvant Hypofractionated Radiotherapy in 15 Versus 5 Fractions After Breast Conserving Surgery or Mastectomy for Early or Locally Advanced Breast Cancer in Women Above 65 Years
Brief Title: Outcome of 15 Versus 5 Fractions in Adjuvant Breast Radiotherapy in Women Over 65 Years
Acronym: HAI-5-III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2016/1386
Record Dates: First submitted 2017-01-13; First posted 2017-04-20 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Breastcancer
Keywords: Accelerated radiotherapy; Older women; Hypo-fractonation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- WBI - randomized - 5 (Experimental): WBI 5 fractions SIB 5 fractions if needed
  Interventions: Radiation: WBI 5 fractions; Radiation: SIB 5 fractions if needed
- WBI - randomized - 15 (Active Comparator): WBI 15 fractions SIB 15 fractions if needed
  Interventions: Radiation: WBI 15 fractions; Radiation: SIB 15 fractions if needed
- WBI - observational - 5 (Experimental): WBI 5 fractions SIB 5 fractions if needed
  Interventions: Radiation: WBI 5 fractions; Radiation: SIB 5 fractions if needed
- WBI - observational - 15 (Active Comparator): WBI 15 fractions SIB 15 fractions if needed
  Interventions: Radiation: WBI 15 fractions; Radiation: SIB 15 fractions if needed
- WBI + LNI - randomized - 5 (Experimental): WBI 5 fractions SIB 5 fractions if needed LNI 5 fractions
  Interventions: Radiation: WBI 5 fractions; Radiation: LNI 5 fractions; Radiation: SIB 5 fractions if needed
- WBI + LNI - randomized - 15 (Active Comparator): WBI 15 fractions SIB 15 fractions if needed LNI 15 fractions
  Interventions: Radiation: WBI 15 fractions; Radiation: LNI 15 fractions; Radiation: SIB 15 fractions if needed
- WBI with LNI - observational - 5 (Experimental): WBI 5 fractions SIB 5 fractions if needed LNI 5 fractions
  Interventions: Radiation: WBI 5 fractions; Radiation: LNI 5 fractions; Radiation: SIB 5 fractions if needed
- WBI with LNI - observational - 15 (Active Comparator): WBI 15 fractions SIB 15 fractions if needed LNI 15 fractions
  Interventions: Radiation: WBI 15 fractions; Radiation: LNI 15 fractions; Radiation: SIB 15 fractions if needed
- thoracic wall irradiation (TWI) +/- LNI - observational - 5 (Experimental): TWI 5 fractions SIB 5 fractions if needed LNI 5 fractions
  Interventions: Radiation: LNI 5 fractions; Radiation: TWI 5 fractions
- TWI +/- LNI - observational - 15 (Active Comparator): TWI 15 fractions SIB 15 fractions if needed LNI 15 fractions
  Interventions: Radiation: LNI 15 fractions; Radiation: TWI 15 fractions

INTERVENTIONS:
Radiation: WBI 5 fractions — External beam radiotherapy in 5 fractions of 5,7Gy
  Arms: WBI + LNI - randomized - 5; WBI - observational - 5; WBI - randomized - 5; WBI with LNI - observational - 5
Radiation: WBI 15 fractions — External beam radiotherapy in 15 fractions of 2,67Gy
  Arms: WBI + LNI - randomized - 15; WBI - observational - 15; WBI - randomized - 15; WBI with LNI - observational - 15
Radiation: LNI 5 fractions — External beam radiotherapy in 5 fractions of 5,4Gy
  Arms: WBI + LNI - randomized - 5; WBI with LNI - observational - 5; thoracic wall irradiation (TWI) +/- LNI - observational - 5
Radiation: LNI 15 fractions — External beam radiotherapy in 15 fractions of 2,67Gy
  Arms: TWI +/- LNI - observational - 15; WBI + LNI - randomized - 15; WBI with LNI - observational - 15
Radiation: SIB 5 fractions if needed — Simultaneous boost of 5 x 6,2Gy (6,5Gy in case of involved resection margins) if needed
  Arms: WBI + LNI - randomized - 5; WBI - observational - 5; WBI - randomized - 5; WBI with LNI - observational - 5
Radiation: SIB 15 fractions if needed — Simultaneous boost of 15x3,12Gy (3,33Gy in case of involved resection margins) if needed
  Arms: WBI + LNI - randomized - 15; WBI - observational - 15; WBI - randomized - 15; WBI with LNI - observational - 15
Radiation: TWI 5 fractions — External beam radiotherapy in 5 fractions of 5,7Gy
  Arms: thoracic wall irradiation (TWI) +/- LNI - observational - 5
Radiation: TWI 15 fractions — External beam radiotherapy in 15 fractions of 2,67Gy
  Arms: TWI +/- LNI - observational - 15

SUMMARY:
This study will evaluate the effect of highly accelerated external beam radiotherapy (EBRT) in 5 fractions over 10 days compared to 15 fractions over 3 weeks for early as well as locally-advanced stage breast cancer.

Primary endpoint will be chronic toxicity (breast deformation and retraction). Secondary endpoints are acute toxicity, loco-regional and distant tumor control, patient reported QoL and cosmetic satisfaction. Patients with lymph node irradiation will be closely monitored for radiation induced plexopathy.

DETAILED DESCRIPTION:
Over the age of 65, uptake of adjuvant radiotherapy after surgery for breast cancer declines, even in women with poor prognostic stage or adverse tumor characteristics.

Lowering the number of fractions may reduce reluctancy for radiotherapy in this age group.

In a preceding prospective phase I-II trial, evaluating EBRT over 10 days, results on technical feasibility and acute toxicity were positively evaluated.

However, data on the chronic effects of breast irradiation using high doses per fraction are still sparse.

This trial is developed to compare standard hypo-fractionation in 15 fractions (if needed with simultaneously integrated boost - SIB) with highly accelerated radiotherapy in 5 fractions.

Patients referred for adjuvant radiotherapy after breast conserving surgery will preferably be randomized, depending on the indication, to a study-arm with whole breast irradiation (WBI) +/- SIB or to a study-arm with WBI+/- SIB and lymph node irradiation (LNI).

If patients after breast conserving surgery (BCS) have a strong preference for 5 or 15 fractions, they will be invited to enter the parallel observational arm (patient preference).

Patients referred for adjuvant radiotherapy after mastectomy +/- LNI accepting to participate, can choose a 5 or 15-fraction schedule. No randomization is foreseen in this last observational group.

ELIGIBILITY:
Inclusion Criteria:

* breast conserving surgery or mastectomy for breast carcinoma
* multidisciplinary decision of adjuvant irradiation
* absence of distant metastases
* informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* History of previous radiation treatment to the same region
* Bilateral breast irradiation
* Life expectancy of less than 2 years
* Planned reconstructive breast surgery
* Condition making toxicity evaluation difficult, e.g. skin disorders, pre-existing brachial plexus injury, …
* Inability to respect constraints on skin, heart, lungs, esophagus, ribs, brachial plexus or any other organ at risk
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits or unlikely to complete the study

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Breast retraction (LENTSOMA) | 2-5 years
  Breast Cancer Conservative treatment.core (BCCT.core) objective measurement

SECONDARY OUTCOMES:
Acute toxicity: number of patients with clinical relevant dermatitis (CTCAE v. 4.0) | 1-8 weeks
  Assessment of grade of dermatitis
Acute toxicity: number of patients with moist desquamation | 1-8 weeks
  CTCAE v. 4.0 (grade 3)
Acute toxicity: number of patients with pain (CTCAE v. 4.0) | 1-8 weeks
  Grade 1: mild; Grade 2: moderate, limiting activity of daily living (ADL); grade 3: severe, limiting ADL
Acute toxicity: number of patients with pruritus (CTCAE v. 4.0) | 1-8 weeks
  Grade 1: mild, localized topical intervention; Grade 2: intense, oral intervention, skin changes
Acute toxicity: number of patients with fatigue (MFI-20) | 1-8 weeks
  Questionnaire (20 questions)
Chronic toxicity: measurement of patient satisfaction with breast esthetic outcome | Before radiotherapy and after 2 and 5 years
  BREAST-Q questionnaire: Patient reported outcome, evaluating satisfaction with esthetic outcome.
Chronic toxicity: prevalence of fibrosis | 2 and 5 years
  LENT Soma: fibrosis (score 0-3)
Chronic toxicity: prevalence of pain | 2 and 5 years
  LENT Soma: score 0-4
Chronic toxicity: prevalence of telangiectasia | 2 and 5 years
  LENT Soma: Score 0-3
Chronic toxicity: prevalence of lymphedema | 2 and 5 years
  LENT Soma: score 0-4
Chronic toxicity: prevalence of fatigue (MFI-20) | 2 and 5 years
  Questionnaire (20 questions)
Chronic toxicity - prevalence of radiation induced brachial plexopathy (RIBP) (standardized screening questionnaire), confirmed by electromyogram (EMG) | 2 and 5 years
  If a screening reveals unilateral pain, loss of function or muscular atrophy in the ipsilateral arm, an EMG will be performed to confirm/exclude RIBP
Loco-regional tumor control | 2 and 5 years
  Ipsilateral or regional breast recurrence
Distant tumor control | 2 and 5 years
  Distant metastases free survival
Breast cancer specific survival | 2 and 5 years
  Number of patients alive and without breast cancer recurrence at 2 and 5 years after adjuvant radiotherapy
Overall survival | 2 and 5 years
  Number of patients alive, 2 and 5 years after adjuvant radiotherapy

OTHER OUTCOMES:
Patient preference | Moment of intake, before allocation to study arm.
  Patients can accept clinical trial but refuse randomization. In this case they will be allocated to a patient preference study arm, existing also of a 5 or 15 fraction-schedule. The choice of the patient: acceptance or non-acceptance of study, acceptance or non-acceptance of randomization, in case of patient preference arm: acceptance or 5 or 15 fractions.
QoL within perspective of cancer patients | 4 weeks, 1, 2 and 5 years
  QLQ C30 - standardised questionnaire
QoL within perspective of breast cancer patients | 4 weeks, 1, 2 and 5 years
  QLQ BR23 - standardised questionnaire
QoL within perspective of healthy patients | 4 weeks, 1, 2 and 5 years
  EQ-D5: standardised questionnaire
Number of patients evolving to higher frailty score after radiotherapy | 4 weeks, 1, 2 and 5 years
  Measurement of frailty using G8 geriatric screening tool
Cost Effectiveness Analysis | 5 years
  Cost effectiveness analysis comparing 5 with 15 fractions
Technical feasibility of prone positioning | At the moment of simulation
  Percentage of patients able to perform prone positioning on new breast board: yes or no.
Technical feasibility of deep inspirational breath-hold in prone position | At the moment of simulation
  Percentage of patients able to perform breath-hold procedure in prone position: yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Liv Veldeman, M.D., PhD, Principal Investigator — Ghent University Hospital, Dept. Radiotherapy-Oncology
Locations (1):
- Ghent University Hospital, Dept. Radiotherapy-Oncology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HAI-5 feasilibility trial: results acute toxicity — http://dx.doi.org/10.1016/j.ijrobp.2017.01.229